CLINICAL TRIAL: NCT00276029
Title: The Efficacy of a Soluble Ligand Binding Tumour Necrosis Factor Receptor, Etanercept, in Severe, Steroid Dependant Asthma: a Randomised Controlled Study
Brief Title: TNF Alpha in Refractory Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: etanercept/pr2
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2006-05-04 (Estimated); Status verified 2004-09

CONDITIONS: Asthma
Keywords: Asthma; Refractory
MeSH Terms: conditions — Asthma | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this study was to investigate whether the administration of etanercept to patients with severe asthma improved their asthma related quality of life and a measure of the degree of reactivity of the airways

DETAILED DESCRIPTION:
Although steroid dependent asthma represents a small population of patients with asthma, they consume a disproportionately large amount of the health resource burden attributed to asthma. Treatment options in this group are extremely limited; the development of effective treatments for this group of patients should be a priority, not only for increasing individual patient quality of life but for long term reduction of health spending.

This randomised, double blind, placebo controlled, cross over trial will investigate the efficacy of a soluble TNF receptor, etanercept, in severe, steroid dependant asthma.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic asthma Methacholine PC20<8mg/ml

Exclusion Criteria:

* History of poor treatment concordance History of tuberculosis Radiographic evidence of previous tuberculosis Recent tuberculosis contact Respiratory tract infection within 3 months Current Smoker or Ex-smoker with more than 5 pack years Symptomatic co-morbid condition Contra-indication to etanercept Pregancy Breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2003-12; Study Completion 2004-09

PRIMARY OUTCOMES:
Methacholine PC20
Juniper asthma quality of life

SECONDARY OUTCOMES:
Net change in post-bronchodilator FEV1
FEF25-75
FVC
symptom visual analogue score
exhaled nitric oxide concentration
computed alveolar nitric oxide concentration
sputum differential inflammatory cell counts
sputum supernatant mediator concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Berry, MB, ChB, Principal Investigator — Institute for Lung Health
Locations (1):
- Institute for Lung Health, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Result] Berry MA, Hargadon B, Shelley M, Parker D, Shaw DE, Green RH, Bradding P, Brightling CE, Wardlaw AJ, Pavord ID. Evidence of a role of tumor necrosis factor alpha in refractory asthma. N Engl J Med. 2006 Feb 16;354(7):697-708. doi: 10.1056/NEJMoa050580. PMID 16481637